CLINICAL TRIAL: NCT00671541
Title: Nasospore Stent For The Use in Endoscopic Sinus Surgery
Brief Title: Nasospore Stent For Use in Enodscopic Sinus Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Principal Investigator left the institution requested study terminated.
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LCID 2006-026
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Sinusitis
MeSH Terms: interventions — Bacitracin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Merogel stent vs. Nasopore Stent (Active Comparator): This study has two arms consiting of 50 subjects each (100 total) Arm 1 will recieve the standard stent (merogel)in their right sinus and a nasopore stent in their left sinus.
  Interventions: Drug: Merogel Nasal Stent and Nasopore Stent
- bacitracin vs. gentamicin treated stent (Experimental): The second arm will consist of 50 new subjects. These 50 subjects will have a nasopore stent placed in the left sinus. The first 25 subjects will have nasopore stent placed postoperatively with a bacitracin soaked nasopore in right sinus the second 25 will have a gentamycin soaked nasopore stent in right sinus.
  Interventions: Drug: Merogel Nasal Stent and Nasopore Stent; Drug: Nasopore Stent and either Gentamycin or Bacitracin

INTERVENTIONS:
Drug: Merogel Nasal Stent and Nasopore Stent — Merogel Nasal Stent and Nasopore Stent
  Other Names: Merogel Stent; Nasopore Stent; Bacatracin soaked stent; Gentamicin soaked stent
Drug: Nasopore Stent and either Gentamycin or Bacitracin — Nasopore Stent with Bacitracin (100,000 units in 10cc(NSS)or Gentamycin(80mg in 10cc NSS)
  Other Names: Merogel Stent; Nasopore Stent; Bacatracin soaked stent; Gentamicin soaked stent
  Arms: bacitracin vs. gentamicin treated stent

SUMMARY:
The purpose of this study is to evaluate a stenting material called Nasopore. This is a synthetic material approved by FDA for use as a stent in postoperative sinus surgery patients. This study will compare the Nasopore stent to other approved stenting materials.

DETAILED DESCRIPTION:
This study will compare other sinus stenting products to the Nasopore stent. The stents will be soaked in antibiotic solutions and be observed for how well they perform. Subjects will have a stent placed in each sinus, stents may be the standard antibiotic saturated materials or the new nasopore material or nasopore stent soaked in antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Evaluation by Otolaryngologist & determined to need endoscopic sinus surgery
* Only subjects with Bilateral disease

Exclusion Criteria:

* Pediatric subjects(under the age of 18)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
This study will evaluate the efficacy of nasopore stent soaked in bacitracin in and one stent soaked in gentaymcin antibiotic solution | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Catalano, MD, Principal Investigator — Lahey Clinic
Locations (1):
- Lahey Clinic, Inc, Burlington, Massachusetts, United States